CLINICAL TRIAL: NCT06876922
Title: Examination of the Effects of Thoracic Mobility Exercises on Balance, Exercise Capacity, Sleep Quality, Pain and Daily Life Activities in Geriatric Individuals
Brief Title: Effects of Thoracic Mobility Exercises in Geriatric Individuals
Acronym: Geriatric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Buket Büyükturan, Associate Professor, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05.10.2023/ 8 / 37
Record Dates: First submitted 2025-03-03; First posted 2025-03-14 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Geriatric
Keywords: Balance; Exercise Capacity; Geriatrics; Thoracic Mobility; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: 28 geriatric individuals aged 65 and over who do not need care were included in our study and were divided into 2 groups as thoracic mobility exercises and Conventional physiotherapy exercises by randomization. The Conventional physiotherapy exercises; While the thoracic mobility exercises group was made to do conventional exercises including warm-up, stretching, strengthening, posture and breathing exercises, in addition to these exercises, thoracic mobility exercises were done. The individuals included in the study were studied for a total of 8 weeks, 1 week for baseline, 1 week for 6 weeks later and 6 weeks for exercise training.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Thoracic mobility exercises group (Experimental): Thoracic mobility exercises Group: Conventional physiotherapy exercises were given to individuals participating in the Thoracic mobility exercises group. Conventional physiotherapy exercises included warm-up, stretching, strengthening, posture and breathing exercises integrated between them. These exercises were performed in 30-40 minute sessions, 3 days a week and for 6 weeks. Thoracic mobility exercises were applied to individuals participating in the study group in addition to conventional physical therapy exercises.
  Interventions: Other: Thoracic mobility exercises Group
- the Conventional physiotherapy exercises group (Active Comparator): Conventional physiotherapy exercises Group: Conventional physiotherapy exercises were given to individuals participating in the Conventional physiotherapy exercises group. Conventional physiotherapy exercises included warm-up, stretching, strengthening, posture and breathing exercises integrated between them. These exercises were performed in 30-40 minute sessions, 3 days a week and for 6 weeks. Use this module to add descriptions of each arm in the study and to list the interventions being studied.
  Interventions: Other: the Conventional physiotherapy exercises Group

INTERVENTIONS:
Other: Thoracic mobility exercises Group — Thoracic mobility exercises Group: Conventional physiotherapy exercises were given to individuals participating in the control group. Conventional physiotherapy exercises included warm-up, stretching, strengthening, posture and breathing exercises integrated between them. These exercises were performed in 30-40 minute sessions, 3 days a week and for 6 weeks. Thoracic mobility exercises were applied to individuals participating in the study group in addition to conventional physical therapy exercises.
  Arms: the Thoracic mobility exercises group
Other: the Conventional physiotherapy exercises Group — the Conventional physiotherapy exercises Group: Conventional physiotherapy exercises were given to individuals participating in the Conventional physiotherapy exercises group. Conventional physiotherapy exercises included warm-up, stretching, strengthening, posture and breathing exercises integrated between them. These exercises were performed in 30-40 minute sessions, 3 days a week and for 6 weeks. Use this module to add descriptions of each arm in the study and to list the interventions being studied.
  Arms: the Conventional physiotherapy exercises group

SUMMARY:
Aging leads to a gradual decline in muscle function and structural changes in the musculoskeletal system, which can affect balance and increase the risk of falls. This study aimed to assess the effects of thoracic mobility exercises on balance, exercise capacity, sleep quality, pain, and daily activities in 28 geriatric individuals (65+ years). Participants were divided into two groups: the Thoracic mobility exercises group performed conventional exercises with additional thoracic mobility exercises, while the Conventional physiotherapy exercises group did not.

DETAILED DESCRIPTION:
Aging is a natural and irreversible process of the human body that involves a gradual decline in physiological, structural and functional activities. the general muscle function in the body decreases, and in this respect, in addition to structural changes in the musculoskeletal system, there are also changes in the internal function of the muscles. This change may cause an increase in the thoracic curvature in the sagittal plane and postural changes, a shift in the center of gravity forward, disrupting balance and increasing the risk of falling. the intervertebral disc spaces narrow, which causes an increase in the kyphosis angle of the spine. Although studies in the literature use thoracic mobility exercises, the investigators found that these studies specifically evaluate effects on respiratory functions. The aim of this study is to examine the effects of thoracic mobility exercises on balance, exercise capacity, sleep quality, pain and daily living activities in geriatric individuals. 28 geriatric individuals aged 65 and over who do not need care were included in this study and were divided into 2 groups as experimental and control by randomization. The Conventional physiotherapy exercises group; While the thoracic mobility exercises group was made to do conventional exercises including warm-up, stretching, strengthening, posture and breathing exercises, in addition to these exercises, thoracic mobility exercises were done. The individuals included in the study were studied for a total of 8 weeks, 1 week for pre-assessment, 1 week for post-assessment and 6 weeks for exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Elderly individuals over the age of 65
* Those who scored at least 24 points on the mini mental test
* Those who did not need care in their daily living activities

Exclusion Criteria:

* Those with uncontrolled Diabetes Mellitus and Hypertension
* Those with severe obesity
* Those who use medications that may increase the risk of falling
* Those with serious auditory and visual problems
* Those with physical and psychological problems affecting physical mobility
* Those who have undergone surgery in the last 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Beck Balance Scale | baseline- 6 weeks later
  Beck Balance Scale is a scale that evaluates balance in the elderly, where some performance tests are applied to evaluate the deterioration in balance function. It is a valid tool used in clinical practice and research for the evaluation of the effectiveness of interventions and quantitative definitions of function. It consists of 14 items that are scored by observing performance. A ruler, stopwatch, step, chair and 15-20 minutes are required for the application. The highest score is 56. 0-20 indicates balance disorder, 21-40 indicates acceptable balance, and 41-56 indicates good balance.
Time Up-Go test | baseline- 6 weeks later
  To perform the Time Up-Go test, the patient rises from a chair, walks at a comfortable and safe pace to a line on the floor three meters away, turns, and sits back in the chair. The test is attempted once to become familiar with the test. If the patient uses a walking aid, they can perform the test with it. A shorter time indicates better functional performance. A test score of ≥13.5 seconds indicates those at high risk of falling in the community setting. However, threshold values reported in the literature range from 10 to 33 seconds

SECONDARY OUTCOMES:
Evaluation of Exercise Capacity | baseline- 6 weeks later
  A 6-minute walk test was used to evaluate the exercise capacity of elderly individuals. The 6MWT is a well-known, valid, and reliable measure of aerobic capacity in elderly people with heart, peripheral vascular, and respiratory diseases. The 6MWT has also been used as an indicator measure of submaximal aerobic capacity in the elderly population. The test should be performed in a flat, hard-surfaced corridor at least 30 meters long. The patient is told to be calm, have taken their medications, and wear comfortable clothes and shoes. Once the patient understands the instructions, they are ready to begin the test. Vital signs are recorded before starting the test. During the test, participants must walk at a pace appropriate to their condition and may stop, slow down, and continue walking as soon as possible if they wish. The therapist may encourage the patient with standard phrases such as 'You're doing well', 'Keep up the good work'. At the end of the test, the therapist measures vita
Evaluation of Sleep Quality | baseline- 6 weeks later
  Pittsburgh Sleep Quality Index (PSQI) was used to test the sleep quality of elderly individuals. PSQI is a 19-item self-report scale that evaluates sleep quality and disturbances in the past month. It consists of 24 questions, 19 of which are self-report questions and 5 of which are questions to be answered by the spouse or roommate. The 18 questions scored on the scale consist of 7 components. Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disturbance, Use of Sleeping Pills and Daytime Dysfunction. Each component is evaluated on a scale of 0-3 points. The total score of the 7 components gives the total scale score. The total score varies between 0-21. A total score greater than 5 indicates "poor sleep quality".
The Geriatric Pain Scale | baseline- 6 weeks later
  The Geriatric Pain Scale was used to assess the pain status of elderly individuals. The scale consists of 5 dimensions: withdrawal due to pain, pain intensity, pain with movement, pain with strenuous activities and pain with other activities. Two items in the scale are included in two sub-dimensions at the same time, and there are also 3 open-ended questions about pain in the scale. 22 items in the scale are scored in binary form, and the other 2 items are scored on a 0-10 scale. The total score is found by adding the "Yes" answers and varies between 0-42. Each item in the scale is converted to the 0-100 system by multiplying it by 2.38. The final score of the scale is calculated by converting it to a 0-100 scale. In the evaluation of the Geriatric Pain Scale, the scores range from 0 to 100, with scor
The Bartel daily life activity assessment scale | baseline- 6 weeks later
  The Bartel daily life activity assessment scale was used to evaluate the daily life activities of the elderly. This scale consists of 10 items that rate the functions of nutrition, washing, self-care, dressing, defecation control, urinary control, going to the toilet, the ability to move from bed to wheelchair, mobility status such as walking or being wheelchair dependent, and climbing stairs on a 5-15 point scale based on increasing difficulty between tasks. The aim of this scale is to determine the patient's level of disability. It is not necessary to test the patient directly, but evaluation can be made in the light of direct observation, information obtained from the patient, the patient's relatives, or the caregiver or nurse involved in their care.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran Univercity, Kırşehir, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I was undecided because I didn't know what the benefit would be to me if I shared it or not.